CLINICAL TRIAL: NCT00738426
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia ML Scanner (MLS) on Body Contouring of the Waist, Hips and Thighs Clinical Study Protocol
Brief Title: Study of Low Level Laser Therapy for Body Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCL-001
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Body Contouring
Keywords: non-invasive body contouring of waists hips and thighs

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia ML Scanner (MLS) (Active Comparator): Red diode low level laser light energy
  Interventions: Device: Erchonia ML Scanner (MLS)
- Sham device (Sham Comparator): non-therapeutic sham light output
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Erchonia ML Scanner (MLS) — Red diode low level laser light energy.
  Arms: Erchonia ML Scanner (MLS)
Device: Sham device — non-therapeutic light energy output
  Arms: Sham device

SUMMARY:
The purpose of this study is to determine whether green diode low level laser therapy is effective for body contouring of the waist, hips and thighs.

DETAILED DESCRIPTION:
Weight loss and body contouring are large, constantly-growing fields of cosmetic surgery. According to the American Society of Plastic Surgeons (ASPS) statistics, more than 324,000 liposuction procedures, 233,000 eyelid surgeries and 114,000 facelift procedures were performed in 2004 in the United States alone. However, while the demand for body shaping procedures is constantly on the rise, so is the demand for such procedures to be performed more quickly, simply and most importantly, less invasively. Cosmetic surgery patients are no longer satisfied with procedures that require general anesthesia, pose a multitude of potentially serious risks and complications and that require several weeks of recovery time. Hence the growing popularity of non- to minimally-invasive cosmetic surgery procedures. In 2005, more than 7.5 million minimally-invasive cosmetic procedures were performed, a 35% increase from 2000. Consequently, patients and physicians alike are continually searching for non-invasive alternatives to traditional cosmetic procedures such as liposuction that are efficient, safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* indicated for liposuction for the removal of localized deposits of adipose tissues that do not respond to diet and exercise; specifically in the areas of the waist, hips and bilateral thighs.
* willing and able to abstain from partaking in any treatment other than the study procedure (existing or new) to promote body contouring and/or weight loss during the course of study participation.
* willing and able to maintain regular diet and exercise regimen without during study participation.
* 18 to 65 years.
* Male or female.

Exclusion Criteria:

* Body Mass Index (BMI) of 30 kg/m² or greater.
* Diabetes dependent on insulin or oral hypoglycemic medications.
* known cardiovascular disease.
* cardiac surgeries, pacemakers.
* excessive alcohol consumption.
* prior surgical intervention for body sculpting/weight loss.
* medical, physical, or other contraindications for body sculpting/weight loss.
* current use of medication(s) known to affect weight levels and/or to cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent.
* medical condition known to affect weight levels and/or to cause bloating or swelling.
* diagnosis of, and/or taking medication for, irritable bowel syndrome.
* active infection, wound or other external trauma to the areas to be treated with the laser.
* pregnant, breast feeding, or planning pregnancy prior to study end.
* serious mental health illness; psychiatric hospitalization in past two years.
* developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to weight-related and/or body shape issues.
* participation in research in the past 90 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Roche, MD, FACS, Principal Investigator; Robert F Jackson, MD, FACS, Principal Investigator
Locations (3):
- United States (3):
  - Douglas D. Dedo, MD, FACS, Palm Beach Gardens, Florida
  - Cosmetic Surgery, Marion, Indiana
  - Dr. Gregory C. Roche, Bloomfield Hills, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia ML Scanner (MLS) | Sham Device
Started | 37 | 35
Completed | 35 | 32
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia ML Scanner (MLS) | Sham Device | Total
Number analyzed (Participants) | 35 | 32 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 34 | 32 | 66
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 32 | 67
  >=65 years | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Reduction of at Least 3.0 Inches Off Their Combined Waist-hips-thighs Circumference.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia ML Scanner (MLS) | Sham Device
Number analyzed (Participants) | 35 | 32
participants | 21 | 2

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Erchonia ML Scanner (MLS) | Sham Device
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No